CLINICAL TRIAL: NCT01121861
Title: Prospective Comparative Study of the Efficacy, Predictability, Safety and Stability of the STAAR and Alcon Toric Intraocular Lenses Implanted in Asian Eyes During Phacoemulsification Surgery
Brief Title: Prospective Comparative Study of Refractive Outcome of STAAR and Alcon Toric Intraocular Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R536/24/2007
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Astigamtism
Keywords: efficacy; safety; predictability; stability; toric IOL; refractive astigmatism; phacoemulsification
MeSH Terms: interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Phacoemulsification with implantation of toric IOL

SUMMARY:
Several methods have been developed to address and reduce preexisting astigmatism. The refractive results associated with the use of toric IOLs are likely to be more predictable. Other advantages of toric IOL include absence of need for any additional astigmatic correction procedure during cataract surgery, faster visual recovery as well as the reversibility of the procedure. There has not been any trial carried out to evaluate the results of toric IOL in either the investigators local population or in East Asia. Hence, the investigators set out to evaluate and compare the efficacy, safety, predictability and stability of the STAAR and Alcon toric IOL in Asian eyes.

DETAILED DESCRIPTION:
The improvements in surgical technique as well as advances in technology employed during modern cataract surgery have made it a safe procedure in routine cases. Moving forwards, the single most pressing challenge facing cataract surgeons in the developed countries today is the ability to achieve predictable and accurate refractive outcomes. Increasingly, surgeons and patients alike have come to measure the success of their surgery by the refractive outcome.

Using partial coherence interferometry has led to more accurate biometry and consequently more predictable spherical results. This also helped paved the way for satisfactory correction of presbyopia with multifocal intraocular lenses (IOL).

Astigmatism is also an important component of the refractive equation. Estimates of the incidence of significant, naturally occurring astigmatism vary widely from 7.5% to 75%1. It is thought that 3% to 15% of eyes may have 2 or more diopters (D) of astigmatism2. Many surgeons would agree that astigmatism of greater than 0.5 D will have visual consequences such as symptoms of ghosting and shadows and they now aim for both spherical and astigmatic outcomes of +/ - 0.5 D3.

Several methods have been developed to address and reduce preexisting astigmatism. While corneal relaxing incisions for astigmatic correction can be unpredictable and highly surgeon dependent, the opposite is true for toric IOLs. The refractive results associated with the use of toric IOLs are likely to be more predictable as it is independent of corneal wound healing. The implantation of an IOL is also less surgeon dependent. Other advantages associated with toric IOLs include the absence of need for any additional astigmatic correction procedure during cataract surgery, faster visual recovery as well as the reversibility of the procedure.

Studies have been carried out to evaluate the efficacy and rotational stability of the STAAR AA4203 TF/TL toric IOL since its FDA approval in November 1998. These trials have only been carried out on Caucasian eyes and have shown a significant reduction in the pre-existing refractive astigmatism, improvement of postoperative unaided visual acuity as well as excellent refractive as well as rotational stability (latter especially so with the TL model). Ruhswurm et al.6 reviewed 37 eyes with STAAR toric IOL over a mean duration of 20.3 months and found that 78.4% of eyes had residual refractive astigmatism within +/- 1.00 D and 48.6% within +/- 0.50D. 83.4% of these eyes achieved best-corrected visual acuity of 20/40 or better. Sun et al.7 demonstrated improved unaided visual outcome between eyes with toric (130 eyes; 86.4% with visual acuity 20/40 or better) and spherical IOL (51 eyes; 76% with visual acuity 20/40 or better). Similar results have also been obtained with the Alcon toric IOL. In Horn et al.9, the clinical trial results of 250 patients with Alcon toric IOL have been described, demonstrating good unaided visual acuity of 20/25 or better at the 6-month postoperative visit (66% of patients with unilateral toric implant and 97% with bilateral implants). 97% of these toric patients achieved spectacle freedom for distance vision, compared to 50% of control patients. It is well documented that the rotational stability of these toric IOL is crucial to the efficacy of astigmatic reduction. Theoretical calculations show that an estimated 1/3 of astigmatic correction is lost if the IOL is rotated by 10 degrees off axis, as well as potential worsening of preoperative astigmatism in the presence of more than 30 degrees of off-axis rotation. Toric IOL stability is dependent on multiple factors, one of which is the capsular bag size. Vass et al.11 showed a good correlation between axial length and capsular bag diameter (CBD), especially so in eyes with axial lengths of less than 25.0mm. On the other hand, highly myopic eyes are not shown to have a greater risk of having a larger CBD than those with normal axial lengths. A formula derived to calculate a predicted CBD (CBDp) showed that values greater than 10.3mm are likely to have existing larger CBD and hence benefit from implantation of longer toric IOL due to better centration.

To date, there has not been any trial carried out to evaluate the results of toric IOL in either our local population or in East Asia. There has also not been any prospective clinical trial conducted to compare the difference (if any) between a plate-haptic and loop-haptic toric IOL. Hence, we set out to evaluate and compare the efficacy, safety, predictability and stability of the STAAR and Alcon toric IOL in Asian eyes.

ELIGIBILITY:
Inclusion Criteria:

1. Suitability for phacoemulsification surgery.
2. Regular corneal astigmatism of at least 1.25D and not exceeding 2.0D.
3. Age range between 21-80 years.
4. Informed consent of surgery and implantation of toric IOL obtained.

Exclusion Criteria:

1. Presence of irregular corneal astigmatism.
2. Regular corneal astigmatism less than 1.0D.
3. Presence of other ocular diseases that may compromise on the visual outcome such as glaucoma, retinal diseases, macular diseases and corneal diseases.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Amount of astigmatism reduction | 3 months

SECONDARY OUTCOMES:
Stability of toric IOL | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wei Han Chua, FRCS, FAMS, Principal Investigator — Singapore National Eye Centre; Jocelyn Chua, MRCS, MMED, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

REFERENCES:
- [Background] Horn JD. Status of toric intraocular lenses. Curr Opin Ophthalmol. 2007 Feb;18(1):58-61. doi: 10.1097/ICU.0b013e328011f9bf. PMID 17159449
- [Result] Till JS, Yoder PR Jr, Wilcox TK, Spielman JL. Toric intraocular lens implantation: 100 consecutive cases. J Cataract Refract Surg. 2002 Feb;28(2):295-301. doi: 10.1016/s0886-3350(01)01035-5. PMID 11821213
- [Result] Chang DF. Early rotational stability of the longer Staar toric intraocular lens: fifty consecutive cases. J Cataract Refract Surg. 2003 May;29(5):935-40. doi: 10.1016/s0886-3350(02)01843-6. PMID 12781279
- [Result] Sun XY, Vicary D, Montgomery P, Griffiths M. Toric intraocular lenses for correcting astigmatism in 130 eyes. Ophthalmology. 2000 Sep;107(9):1776-81; discussion 1781-2. doi: 10.1016/s0161-6420(00)00266-9. PMID 10964844
- [Result] Patel CK, Ormonde S, Rosen PH, Bron AJ. Postoperative intraocular lens rotation: a randomized comparison of plate and loop haptic implants. Ophthalmology. 1999 Nov;106(11):2190-5; discussion 2196. doi: 10.1016/S0161-6420(99)90504-3. PMID 10571358